CLINICAL TRIAL: NCT04604678
Title: Pilot Study Into the Use of Metformin and Low Dose Naltrexone (LDN) for Patients With Coronavirus Disease 2019 (COVID-19) - Assessment of Short and Long Term Effects
Brief Title: Pilot Study Into the Use of Metformin and LDN for Patients With COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit participants due to restrictive inclusion/exclusion criteria. Will update protocol with IRB & begin anew after approval.
Sponsor: AgelessRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALRx003
Record Dates: First submitted 2020-10-26; First posted 2020-10-27 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Covid19
Keywords: metformin; LDN; low dose naltrexone; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Metformin; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Metformin and LDN (Experimental): Patients will be treated with 1500 mg/day of metformin and 4.5 mg/day of LDN for a total of 4 weeks.
  Interventions: Drug: Metformin; Drug: Naltrexone
- Regular health care comparison group (No Intervention): Patients will receive regular health care and will serve as a control group.

INTERVENTIONS:
Drug: Metformin — Metformin at 1500 mg/day
  Arms: Treatment with Metformin and LDN
Drug: Naltrexone — Naltrexone at 4.5 mg/day (LDN)
  Other Names: LDN
  Arms: Treatment with Metformin and LDN

SUMMARY:
Study into the effects of daily use of metformin and low-dose naltrexone (LDN) for 4 weeks to reduce symptoms, disease severity, and recovery time from COVID-19.

DETAILED DESCRIPTION:
The researchers will treat 40 patients with metformin (1500 mg/day) and LDN (4.5 mg/day) for 4 weeks to reduce symptoms, disease severity, and recovery time from COVID-19. These 40 patients will be compared with 40 control patients who will receive regular care. All patients will be asked to complete surveys at baseline and after 1, 2, and 4 weeks after initiation of treatment. The difference with baseline at each time point will be assessed. The surveys will assess COVID-19 symptoms severity.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-70
* Any sex
* Any ethnicity
* Adequate cognitive function to be able to give informed consent
* Technologically competent to complete web forms and perform video calls with the PI
* Positive PCR (polymerase chain reaction) test result for SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) within the last 10 days
* At least two COVID-19 symptoms as assessed by laboratory or patient self-reporting started within the last 3 days
* Willing to fill out regular questionnaires
* Willing to take metformin and LDN

Exclusion Criteria:

* Clinically significant hepatic, renal, or cardiac impairment (as determined by previous clinical judgement)
* Hypoglycemia
* Currently on drugs for COVID-19
* Hospitalization for COVID-19
* (Suspected) pregnancy or breastfeeding
* Active cancer
* Uncontrolled mental health issues
* On any medication with major interactions with metformin or LDN
* Taking opioid analgesics, or being treated for opioid addiction/recovery
* Opioid dependence or withdrawal syndrome
* Known sensitivity to metformin or naltrexone
* Current users of metformin or naltrexone

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of COVID-19 symptoms after 1 week of treatment with metformin and LDN | 1 week
  Reduction in COVID-19 symptoms as measured with the COVID-19 Symptoms Severity Scale. The scale has a minimum score of 0 and a maximum of 24, with values ranging from 4-11 are considered 'mild symptoms', scores ranging 12-19 are considered 'moderate', and scores 20-24 are considered 'severe'.
Reduction of COVID-19 symptoms after 2 weeks of treatment with metformin and LDN | 2 weeks
  Reduction in COVID-19 symptoms as measured with the COVID-19 Symptoms Severity Scale. The scale has a minimum score of 0 and a maximum of 24, with values ranging from 4-11 are considered 'mild symptoms', scores ranging 12-19 are considered 'moderate', and scores 20-24 are considered 'severe'.

SECONDARY OUTCOMES:
Reduction in recovery time from COVID-19 | 4 weeks
  Reduction in the number of days with symptoms due to COVID-19 upon treatment with metformin and LDN, compared to placebo group
Reduction in hospitalizations | 4 weeks
  Reduction in the number of patients being hospitalized due to COVID-19 upon treatment with metformin and LDN, compared to placebo group
Reduction in requirement of additional treatment due to COVID-19 | 4 weeks
  Reduction in the number of patients requiring additional treatment for COVID-19 upon treatment with metformin and LDN, compared to placebo group
Reduction in mortality | 4 weeks
  Reduction in the number of mortality cases due to COVID-19 upon treatment with metformin and LDN, compared to placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Sajad Zalzala, MD, Study Director — AgelessRx; Sajad Zalzala, MD, Principal Investigator — AgelessRx
Locations (1):
- AgelessRx, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No